CLINICAL TRIAL: NCT04878809
Title: Rapid Screening Circuit of COVID 19 in Schools, Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación FLS de Lucha Contra el Sida, las Enfermedades Infecciosas y la Promoción de la Salud y la Ciencia (Other)
Collaborators: Escola L'Horitzó (Unknown); Escola John Talabot (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ESCORAT
Record Dates: First submitted 2021-04-28; First posted 2021-05-07 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-06

CONDITIONS: SARS-CoV-2 (COVID-19)
Keywords: SARS-CoV-2; COVID-19; Coronavirus; School
MeSH Terms: conditions — COVID-19; Coronavirus Infections

STUDY DESIGN:
Intervention Model Description: Experimental Group: People attending L'Horitzó School (students, teachers, administrative and service staff) Control Group (No Intervention): Escola John Talabot
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): People attending L'Horitzó School (students, teachers, administrative and service staff)
  Interventions: Other: Escola L'Horitzó
- Control Group (Other): Escola John Talabot, will provide the incidence rate of infections by SARS-CoV-2
  Interventions: Other: Escola John Talabot

INTERVENTIONS:
Other: Escola L'Horitzó — Diagnosis of SARS-CoV-2 infection by rapid antigen detection tests in nasal and nasopharyngeal swabs, in asymptomatic and symptomatic subjects who attend regularly to L'Horitzó school .
  Arms: Experimental group
Other: Escola John Talabot — John Talabot School will provide the incidence of infection by SARS-CoV-2 in order to compare the incidence of infection from L'Horitzó School.
  Arms: Control Group

SUMMARY:
The outbreak of coronavirus disease 2019 (COVID-19), caused by acute respiratory syndrome severe coronavirus 2 (SARS-CoV-2), emerged in Wuhan in December 2019 and has spread which poses a serious threat to public health. While 80% of the patients are asymptomatic or have a mild illness, 20% develop a serious illness. Predominant symptoms include fever, cough, and myalgias.

Most children have one mild or asymptomatic disease that can be resolved without medical attention and that, exceptionally, may progress to pneumonia and respiratory failure requiring hospitalization

Schools have started the course with strict protocols to prevent the transmission of SARS-Cov-2 among the members of the educational communities and thus avoid an uncontrollability of the epidemic. These protocols include scaled entrances in the centers and differentiated circulation to optimize compliance with social distance. They also include the creation of coexistence groups, the Ventilation of the spaces, hand washing, disinfection of furniture, and wearing a face mask. One key point in the prevention of infection is the rapid detection of infected individuals, their isolation immediate and quarantine, and screening of coexistence groups of positive cases. The diagnosis of Suspicious cases from both schools and other settings is done with a PCR, mostly in Primary Care Centers (PCC). This is causing an increased considerable volume of work for primary care centers.

In addition to the overload of the PCCs, the waiting time between sampling and PCR means that the person must remain at home until the result is obtained, with the negative impact that this means on the daily lives of students, teachers, and families. The use of a quick test performed on the own schools and with staff from the center itself trained to do this first screening would have three very relevant consequences for the system:

1. Speed up the diagnosis and minimize the waiting time between the presentation of symptoms and quarantine of the whole group (if positive)
2. Avoid a waiting time at home with the alteration - often unnecessary - of the day of students, their families, and school staff.
3. Decongest the PCCs, receiving only the cases that need confirmation

DETAILED DESCRIPTION:
The outbreak of coronavirus disease 2019 (COVID-19), caused by acute respiratory syndrome severe coronavirus 2 (SARS-CoV-2), emerged in Wuhan in December 2019 and has spread which poses a serious threat to public health. While 80% of the patients are asymptomatic or have a mild illness, 20% develop a serious illness. Predominant symptoms include fever, cough, and myalgias.

Most children have one mild or asymptomatic disease that can be resolved without medical attention and that, exceptionally, may progress to pneumonia and respiratory failure requiring hospitalization

Schools have started the course with strict protocols to prevent the transmission of SARS-Cov-2 among the members of the educational communities and thus avoid an uncontrollability of the epidemic. These protocols include scaled entrances in the centers and differentiated circulation to optimize compliance with social distance. They also include the creation of coexistence groups, the Ventilation of the spaces, hand washing, disinfection of furniture, and wearing a face mask. One key point in the prevention of infection is the rapid detection of infected individuals, their isolation immediate and quarantine, and screening of coexistence groups of positive cases. The diagnosis of Suspicious cases from both schools and other settings is done with a PCR, mostly in Primary Care Centers (PCC). This is causing an increased considerable volume of work for primary care centers.

In addition to the overload of the PCCs, the waiting time between sampling and PCR means that the person must remain at home until the result is obtained, with the negative impact that this means on the daily lives of students, teachers, and families. The use of a quick test performed on the own schools and with staff from the center itself trained to do this first screening would have three very relevant consequences for the system:

1. Speed up the diagnosis and minimize the waiting time between the presentation of symptoms and quarantine of the whole group (if positive)
2. Avoid a waiting time at home with the alteration - often unnecessary - of the day of students, their families, and school staff.
3. Decongest the PCCs, receiving only the cases that need confirmation

ELIGIBILITY:
Inclusion Criteria:

* Students older than 6 years, teachers, administrative and service staff who attend regularly to L'Horitzó school.
* All participants will be required to sign an informed consent form performing a nasal and nasopharyngeal swab for performing a rapid detection test of antigens (In students under the age of 12, informed consent will be signed by their parent or legal tutor, in students equal to or older than 12 years, but under 18 consent it will be signed both by the student and by his / her parent or legal guardian. The participant over the age of 18 will sign the document in person, unless it is incapacitated, in which case you must sign your legal representative).

Exclusion Criteria:

• Not applicable

Ages: 6 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2021-04-22 (Actual); Primary Completion 2021-06-17 (Actual); Study Completion 2021-06-17 (Actual)

PRIMARY OUTCOMES:
Incidence rate of people infected with SARS-CoV-2 | up to 8 weeks
  Incidence rate of asymptomatic people infected with SARS-CoV-2, detected by rapid antigen detection tests in nasal swabs (self -taken)
Incidence rate of people infected with SARS-CoV-2 | up to 8 weeks
  Incidence rate of symptomatic/asymptomatic people infected with SARS-CoV-2, detected by rapid antigen detection tests in nasopharyngeal swabs performed by trained teachers from the school L'Horitzó

SECONDARY OUTCOMES:
Incidence rate of people infected with SARS-CoV-2 | up to 8 weeks
  Incidence rate of symptomatic people infected with SARS-CoV-2, detected by PCR nasopharyngeal performed under clinical practice.

CONTACTS AND LOCATIONS:
Overall Officials: Boris Revollo Barriga, PhD, MD, Principal Investigator — Fundació FLS de Lluita contra la Sida, les Malalties Infeccioses i la Promoció de la Salut i La Ciència
Locations (2):
- Spain (2):
  - John Talabot, Barcelona
  - Escola l'Horitzó, Barcelona

REFERENCES:
- [Derived] Constantin AM, Noertjojo K, Sommer I, Pizarro AB, Persad E, Durao S, Nussbaumer-Streit B, McElvenny DM, Rhodes S, Martin C, Sampson O, Jorgensen KJ, Bruschettini M. Workplace interventions to reduce the risk of SARS-CoV-2 infection outside of healthcare settings. Cochrane Database Syst Rev. 2024 Apr 10;4(4):CD015112. doi: 10.1002/14651858.CD015112.pub3. PMID 38597249
- [Derived] Pizarro AB, Persad E, Durao S, Nussbaumer-Streit B, Engela-Volker JS, McElvenny D, Rhodes S, Stocking K, Fletcher T, Martin C, Noertjojo K, Sampson O, Verbeek JH, Jorgensen KJ, Bruschettini M. Workplace interventions to reduce the risk of SARS-CoV-2 infection outside of healthcare settings. Cochrane Database Syst Rev. 2022 May 6;5(5):CD015112. doi: 10.1002/14651858.CD015112.pub2. PMID 35514111